CLINICAL TRIAL: NCT06941298
Title: Neural and Psychiatric Consequences of Cannabis Use in Adolescents
Acronym: Cann-Teen
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Nathan Kline Institute for Psychiatric Research (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Vilma Gabbay, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20241204; R01DA059527 (NIH)
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Cannabis Use; Depression
Keywords: Adolescents; Neuroimaging; Functional Magnetic Resonance Imaging (fMRI); Reward; Reward Flanker Task; Reward Predication Error Task; Pain
MeSH Terms: conditions — Depression; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuroimaging Investigation Group (Experimental): Participants in this group will receive neuroimaging investigation for up to 2 years.
  Interventions: Behavioral: Neuroimaging Investigation

INTERVENTIONS:
Behavioral: Neuroimaging Investigation — Participants will undergo fMRI neuroimaging at two timepoints, at the start of the study and at the 1 year follow up. The fMRI is one hour in duration. During the fMRI, participants will complete two tasks investigating diverse aspects of reward circuitry activity. After this is completed, participants will be followed up for another year clinically.

SUMMARY:
The goal of this study is to investigate the effects of cannabis on brain function among adolescents with depression.

ELIGIBILITY:
Inclusion Criteria:

Cannabis users 1) the study team will require majority of adolescents with cannabis use to have a significant cannabis use (self-reported use on ≥15 of the prior 30 days and positive tetrahydrocannabinol (THC) urine toxicology).

Depression Positive

1) participants with subthreshold depression, defined as a raw severity score of ≥30 on the Children's Depression Rating Scale-Revised (CDRS-R, for ages 14-17) and as a raw severity score of ≥12 on the Montgomery Asberg Depression Rating Scale (MADRS, for ages 18-20)

Exclusion Criteria:

1. MRI contraindications such as claustrophobia, metallic ink tattoos, orthodontic braces, or pacemakers
2. positive pregnancy tests
3. neurological illnesses and medical conditions such as unique pain syndromes (e.g. multiple sclerosis, rheumatoid arthritis)
4. estimated full-scale Intelligence Quotient (IQ) ≤80 to ensure that participants have the ability to understand the study112
5. current Substance Use Disorder (SUD) other than cannabis or nicotine.
6. certified for or self-reported medical cannabis use, or intent to become certified
7. current stimulant use (methamphetamine or cocaine) by self-report or urine toxicology
8. oral contraceptives will be allowed and controlled for in order to maximize recruitment of older adolescents.

Depressed THC non-users:

1. psychotropic medication-free for >1 month (or >3 months for medications with a long half- life such as fluoxetine) prior to study enrollment.
2. Diagnostic and Statistical Manual 5 (DSM-5) diagnoses of bipolar disorder, psychotic disorders, autism spectrum all non-cannabis substance-related disorders will be exclusionary.
3. Self-injurious acts (e.g. cutting) and suicidal ideations (SI) without a specific as passive SI) are common in adolescent depression and will be allowed. constitutes an imminent risk to self or others (defined as active SI), the withdrawn from the study and emergency procedures will be initiated immediately,

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Depression Severity measured by the Beck Depression Inventory (BDI) | Up to 3 years
  Scores range from 0-63 with a higher score indicating higher depression severity
Anhedonia Severity measured by the Temporal Experience of Pleasure Scale (TEPS) | Up to 3 years
  Scores range from 18-108 with a higher score indicating higher Anhedonia severity
Cannabis Use measured by the Daily Frequency, Age of Onset, and Quantity of Cannabis Use (DFAQCU) Inventory | Up to 3 years
  Scores range from 1-15 with a higher score indicating more Cannabis Use

SECONDARY OUTCOMES:
Depression Severity measured by the Montgomery-Åsberg Depression Rating Scale (MADRS) | Up to 3 years
  Scores range from 0-60 with a higher score indicating higher depression severity
Depression Severity measured by the Convergence of Children's Depression Rating Scale-revised (CDRSR) | Up to 3 years
  Scores range from 17-113 with a higher score indicating higher depression severity
Anhedonia Severity measured by the Snaith-Hamilton Pleasure Scale (SHAPS) | Up to 3 years
  Scores range from 0-14 with a higher score indicating higher Anhedonia severity
Cannabis Use measured by the Cannabis Use Problems Identification Test (CUPIT) | Up to 3 years
  Scores range from 0-18 with a higher score indicating more Cannabis Use
Cannabis Use measured by a quantitative cannabinoid metabolites urine analysis | Up to 3 years
  will be measured in microgram per liter

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Gabbay, MD, JD, MS, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami Clinical Research Building, Miami, Florida
  - Nathan Kline Institute, Orangeburg, New York

IPD SHARING:
Plan to Share IPD: No